CLINICAL TRIAL: NCT05972005
Title: Stronger At Home: Improve Functional Outcomes for Community-dwelling Older Adults After Hip Fracture
Brief Title: Stronger At Home: Improving Outcomes for Older Adults After Hip Fracture
Acronym: S@H
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Mohammad Auais, PhD (Other)
Responsible Party: Sponsor-Investigator, Dr. Mohammad Auais, PhD, Associate Professor, School Of Rehabilitation Therapy, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6032153
Record Dates: First submitted 2023-07-13; First posted 2023-08-02 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Hip Fractures
Keywords: Hip Fracture; Exercise program; Recovery; Physical therapy
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial (RCT) will be conducted over a period of 14 weeks, utilizing a parallel-group design. It will be a single-blind trial, meaning that the assessors will not be aware of participants assigned intervention. The trial will include repeated measures, with follow-ups conducted up to 12 months after the participants are discharged from the hospital.
  In terms of its design, this trial is considered to be rather pragmatic to very pragmatic, as indicated by a score of 37 out of 45 on the PRECISE-2 tool. The PRECISE-2 tool is used to assess the level of pragmatism in clinical trials, helping to identify trials that closely resemble real-world conditions and are applicable to everyday practice.
Who Masked: Outcomes Assessor
Masking Description: In this type of trial, the researchers responsible for assessing the outcomes remain unaware of the treatment assignments. The purpose of single-blind masking is to minimize bias and ensure that the assessment of outcomes is not influenced by researchers' expectations or knowledge of the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Stronger at Home model) (Experimental): This study implements a 14-week home-based rehabilitation program for older adults after hip fractures. Participants will receive 8 home visits by a Physiotherapist (PT) and/or Physio assistant(PTA), focusing on individualized exercise programs and pain self-management. The intervention aims to improve functional recovery and includes PT-led assessments, exercise adjustments, and discharge assessments. PTAs support exercise delivery and education. The clinical team comprises PTs and PTAs, receiving training on exercise principles, pain education, and goal setting. The program emphasizes progressive strengthening, balance, and functional exercises, adhering to evidence-based principles. The intervention aims to enhance efficiency, reduce wait times, and promote adherence.
  Interventions: Other: The Intervention (Stronger at Home Intervention)
- Control (usual care) (Active Comparator): The control group will receive usual home care provided by the healthcare system, which could vary between cases. We'll document their received care during follow-ups as it is inconsistent and poorly recorded. Regular check-in calls by the study coordinator will remind them of assessments, reducing attrition.
  Interventions: Other: Usual care (Control)

INTERVENTIONS:
Other: The Intervention (Stronger at Home Intervention) — The home-based intervention includes 8 visits by a PT and/or PTA. The PT conducts 3 visits for initial assessment, program design, coaching, and discharge assessments. The program targets personal goals and provides pain self-management support. The second PT visit at 6 weeks allows for reassessment and adjustments. The intervention ensures adherence through multiple sessions, tailored exercises, barrier-solving support, and motivational strategies. The PTA conducts solo visits every other week, assisting with exercises and education under PT supervision. This inclusion reduces wait times and improves efficiency. The clinical team consists of at least 2 PTs and 2 PTAs trained for 3 days. The exercise program adheres to evidence-based principles, involving a 30-minute session with warm-up, exercise, and cool-down. Participants are encouraged to exercise 5 times a week, focusing on strengthening, balance, and functionality. Feasible compliance rates were observed in the pilot study.
  Other Names: The Stronger at Home Physical Therapy program
  Arms: Intervention (Stronger at Home model)
Other: Usual care (Control) — The control group will receive usual home care provided by the healthcare system, which could vary between cases. We'll document their received care during follow-ups as it is inconsistent and poorly recorded. Regular check-in calls by the study coordinator will remind them of assessments, reducing attrition.
  Arms: Control (usual care)

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of a new 14-week individually-tailored home-based rehabilitation program called "Stronger at Home" with usual care in improving functional recovery in community-dwelling older adults after hip fractures.

The main question this trial aims to answer are:

• Is the Stronger at Home program more effective than usual care in improving functional recovery at the end of the 14-week intervention?

secondary questions include:

* What is the cost-utility of the Stronger at Home program compared to usual care at 3.5 months, 6 months, and 12 months after discharge?
* Does the program have a sustained impact on functional recovery at 6 months and 12 months post-discharge?

Participants in the trial will be asked to engage in the following tasks:

* Participate in the Stronger at Home program, which includes using a self-directed toolkit consisting of educational resources and an illustrated exercise program.
* Follow the guidelines provided in the toolkit for gradually increasing exercise intensity and incorporating different types of exercises into their daily life.

The effects of the Stronger at Home program will be compared to those of usual care.

DETAILED DESCRIPTION:
The primary research question of this project is whether the Stronger at Home program, a 14-week individually-tailored home-based rehabilitation program, is more effective than usual care in improving functional recovery in community-dwelling older adults after hip fractures. The evaluation of effectiveness will be conducted at the end of the intervention, which is the primary time point.

In addition to the main research question, secondary aims of the project include evaluating the cost-utility of the Stronger at Home program compared to usual care at 3.5 months, 6 months, and 12 months after discharge. The program's impact on functional recovery will also be assessed at medium-term (6 months) and long-term (12 months) follow-ups after the participants are discharged from the hospital to their homes.

The need for conducting this trial arises from a knowledge gap in effective rehabilitation programs for community-dwelling individuals with hip fractures. The Stronger at Home program was developed through a multistage study incorporating a self-directed toolkit and a new model of care. The development process involved critical analysis of previous programs, adherence to four principles of a successful program, and consultations with researchers, policymakers, older adults, and clinicians. The toolkit includes an educational component and an illustrated exercise program with progressively increasing intensity.

The pilot study of the Stronger at Home program has shown feasibility, with positive feedback from healthcare providers and patients regarding its value.

ELIGIBILITY:
Inclusion Criteria:

* Hip fracture patients who are 55 years or older,
* Currently living in the community, and
* Either being discharged to their home or a retirement home
* Fall from a standing height or less
* Live within 45km radius of recruitment site

Exclusion Criteria:

* Came from long term care or discharged to long term care
* Not a hip fracture (e.g., pelvic fracture)
* Unable to give consent and no proxy
* Fracture due to pathological disease (e.g., cancer, Paget's disease).
* Does not speak English and no translator
* Fracture sustained at hospital
* Terminal illness or exercise contraindications
* Discharged with other services not eligible

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2027-10-17 (Estimated); Study Completion 2028-07-29 (Estimated)

PRIMARY OUTCOMES:
The Lower Extremity Functional Scale (LEFS) | 3.5 months (post intervention )
  The primary outcome of the study (functional abilities) will be assessed using the Lower Extremity Functional Scale (LEFS), a patient-reported outcome measure consisting of 20 items. The LEFS has been validated for various populations, including patients recovering from hip surgeries, and has shown excellent reliability, validity, and responsiveness. It provides a score ranging from 0 to 80 based on the responses to each item's options. The LEFS was chosen based on its ability to evaluate important functional activities for patients, and its use as a primary outcome in the pilot study helped determine the sample size for this trial.

SECONDARY OUTCOMES:
The Short Physical Performance Battery (SPPB) | Baseline, and at 3.5 months, 6 months, and 12 months after discharge.
  The Short Physical Performance Battery (SPPB) will be used as a secondary measure of physical function. The SPPB is a performance-based assessment that includes three tests: standing balance, gait speed, and chair-rising. The total score ranges from 0 to 12, with higher scores indicating better lower extremity physical performance. The SPPB has been extensively validated and used in geriatric research.
Modified Falls Efficacy Scale | Baseline, and 3.5 months, 4.5 months, 6 months, 7.5 months, 9 months, 10.5 months, and 12 months after discharge.
  The Modified Falls Efficacy Scale (MFES) is a commonly used self-report measure designed to assess an individual's confidence in their ability to perform daily activities without falling. It evaluates balance confidence and fear of falling in older adults or individuals with balance impairments. The scale consists of various activities or situations in which falls may occur, and respondents rate their level of confidence in performing each task without falling.
  The MFES typically consists of 14 or 16 items, and each item is rated on a scale ranging from 0% (no confidence) to 100% (complete confidence). The items cover a wide range of activities, including both basic and more complex tasks such as walking on various surfaces, climbing stairs, reaching overhead, and getting out of a chair.
Pain measured with Numerical Analogue Scale (NAS) | Baseline, and 3.5 months, 4.5 months, 6 months, 7.5 months, 9 months, 10.5 months, and 12 months after discharge.
  The NAS will be utilized to assess pain intensity. Participants will be asked to rate their pain levels at rest and during walking on a scale ranging from 0 to 10, with higher scores indicating greater pain intensity.
Tampa Scale of Kinesiophobia (TSK) | Baseline, and 3.5 months, 4.5 months, 6 months, 7.5 months, 9 months, 10.5 months, and 12 months after discharge.
  The TSK will be employed to measure pain-related fear. It assesses individuals' fear and avoidance of physical activity due to pain and provides insights into how fear influences their functional recovery.
2-Minute Walk Test (2MWT) | Baseline, and at 3.5 months, 6 months, and 12 months after discharge.
  The 2MWT will be conducted to evaluate participants' mobility endurance. It measures the distance covered by participants during a 2-minute walk, providing information about their aerobic capacity and endurance.
Clinical Frailty Scale | Baseline and 3.5 months, 6 months, 12 months after discharge
  A summary of the overall level of fitness and/or frailty. Scale of 1-9, with higher scores indicating higher degree of frailty.
Short Depression Scale | Baseline, and 4.5 months, 7.5 months, 9 months, and 10.5 months after discharge
  A 10-item questionnaire related to feelings of depression in the last week.
Short Fear of Falling Scale | Baseline, and 3.5 months, 4.5 months, 6 months, 7.5 months, 9 months, 10.5 months, and 12 months after discharge.
  Scale used to assess fear of falling, with higher scores indicating greater fear of falling

OTHER OUTCOMES:
Health-Related Quality of Life (HRQL) | Baseline, and 3.5 months, 4.5 months, 6 months, 7.5 months, 9 months, 10.5 months, and 12 months after discharge.
  HRQL refers to the impact of a health condition or intervention on a person's well-being. In this study, HRQL will be measured using the EQ-5D. EQ-5D is a generic instrument assessing HRQL across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has three levels (1 = no problems, 2 = some problems, 3 = severe problems).
Quality-Adjusted Life Years (QALYs) | within 7 days of discharge, as well as within 3.5 months, 6 months, 9 months, and 12 months.
  QALYs are a measure of the quantity and quality of life lived. They combine information on HRQL and life expectancy to provide a single summary measure of health outcomes. QALYs will be calculated by assigning utility weights to the HRQL scores obtained from participants and multiplying them by the time spent in that health state.The measurement scale for QALYs ranges from 0 to 1, where 0 represents death and 1 represents perfect health. QALYs are calculated by multiplying the utility weight assigned to a specific health state (obtained from HRQL measures) by the time spent in that state.
Charlson Comorbidity Index | Baseline
  Index developed to capture comorbidities and will be used at baseline to describe the population. Higher scores indicate greater comorbidity.
Sociodemographic information | Baseline
  Survey questionnaire related to living status, employment, smoking status, alcohol consumption, height and weight, income, falls history.
Health Resource Utilization Questionnaire (adapted version) | Baseline, and 3.5 months, 4.5 months, 6 months, 7.5 months, 9 months, 10.5 months, and 12 months after discharge.
  Questionnaire used to capture health utilization. Collects information related to the following: health professional visits, hospital stays, tests/investigations, medications taken, equipment used, access to community resources, time off work, need for paid assistance.
Health Resource Utilization diary | Baseline; 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 months after enrollment.
  Short questionnaire to facilitate data collection for the Health Resource Utilization Questionnaire. Monthly diary sent to participants to record medical appointments, hospital visits, tests, and medications.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No